CLINICAL TRIAL: NCT02376764
Title: New Biomarkers in Post Thrombotic Syndrome
Brief Title: Biomarkers in Post Thrombotic Syndrome
Acronym: BIPOSTO
Status: Completed | Type: Observational
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Prof. Raffaele Serra, University of Catanzaro
Other Study IDs: ER.ALL.2014.04.A
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Postthrombotic Syndrome With Ulcer of Left Lower Extremity; Extracellular Matrix Alteration
MeSH Terms: interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Blood drawing (venipuncture) — Patients with Deep Vein Thrombosis will undergo blood drawing in order to collect plasma samples.

SUMMARY:
This study aims to deepen the investigators knowledge of Post Thrombotic Syndrome and MMPs (and other related molecules such as TIMPS, NGAL and cytokines) to find a predictive molecular system to better classify the risk of patients to develop a PTS after a DVT episode, in order to monitorate more strictly the patients at high risk for developing this complication.

DETAILED DESCRIPTION:
Post-thrombotic syndrome (PTS) is a problem that can develop in nearly half of all patients who experience a deep vein thrombosis (DVT) of lower limbs. PTS symptoms include chronic leg pain, swelling, redness, and skin ulcers. PTS lowers patients' quality of life after DVT, specifically with regards to physical and psychological symptoms and limitations in daily activities. Secondly, the treatment of PTS adds significantly to the cost of treating DVT. PTS also causes lost work productivity: patients with severe PTS and venous ulcers lose up to 2 work days per year Nowadays, there are no effective measures to reduces significatively PTS onset following a DVT episode.

Biomarkers can be of use in further exploring the etiology as well as in developing risk stratification tools for PTS. The relationship between PTS and specific biomarkers may help guide prevention and therapy based on a patient's individual risk profile.

Recent studies showed that MMPs play a significant role in vascular remodeling and endothelial dysfunction and they may explain a role in aneurysm formation as well as in all the clinical manifestations of venous disease (both for acute and chronic related events) but the cellular and molecular mechanisms involved in thrombus resolution and vein wall fibrosis remain undefined.

The presence of MMPs and TIMPs in acute venous occlusion model suggests that there is an important early interplay between protease and inhibitor during events that precede the development of venous disease.

This study aims to deepen the investigators knowledge of PTS and MMPs (and other related molecules such as NGAL and cytokines) to find a predictive molecular system to better classify the risk of patients to develop a PTS after a DVT episode, in order to monitorate more strictly the patients at high risk for developing this complication.

Patients will be recruited at their first episode of DVT and will be followed up according to standard protocols for DVT at 1,4,8,12,24, 36 months. At each visit blood sample will be collected from venipuncture in order to evaluate MMPs (and other related molecules) plasma levels.

These data will be related to clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* Acute DVT of lower limbs.
* no known prior history of DVT
* availability to make follow-up appointments.

Exclusion Criteria:

* prior history of DVT
* neoplasia
* arterial aneurysms
* venous ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Deep Vein Thrombosis of lower limbs during their first episode.
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2012-02; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of plasma MMPs levels | 36 months
  MMPs plasma levels and other related molecules (TIMPS, NGAL and cytokines) will be evaluated during follow up.